CLINICAL TRIAL: NCT00210210
Title: Effect of Ketamine, at the Induction and Its Maintenance to Prevent the Post-operative Pain: Clinical Trial in Cancerology
Brief Title: Administration of Ketamine to Prevent the Post-operative Pain
Acronym: KETAMINE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Institut Bergonié (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IB2004-04; KETAMINE (Other: Institut Bergonié)
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Results first posted 2025-09-08 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Postoperative Pain; Breast Cancer
Keywords: Post-operative-pain; Breast cancer; Morphine; Analgesia
MeSH Terms: conditions — Pain, Postoperative; Breast Neoplasms; Agnosia | interventions — Ketamine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (2):
- Ketamine Arm (Experimental): Anesthetic induction: Ketamine at 0.15 mg/kg is added to the "Reference protocol".
  Anesthetic maintenance: Ketamine at 2 mg/kg/min is added to the "Reference protocol".
  Interventions: Drug: Ketamine
- Reference Arm (Sham Comparator): Induction and anesthetic maintenance without ketamine (reference arm / saline solution)
  Interventions: Drug: Saline solution

INTERVENTIONS:
Drug: Ketamine
  Arms: Ketamine Arm
Drug: Saline solution
  Arms: Reference Arm

SUMMARY:
The surgery of breast cancer is responsible for post-operative pain, needing in about 30% some morphine consumption; like that, the association of ketamine with general anaesthesia may decrease morphine's use and so its adverse effects. The purpose is to evaluate the analgesic effect of a receptor NMDA's antagonist ( ketamine)

ELIGIBILITY:
Inclusion criteria:

* Patients 18 years older
* ASA class 1 or 2
* with surgery of breast cancer (mastectomy or tumorectomy)

Exclusion criteria:

.Kétamine hypersensitivity

* Major psychiatric disorders
* Major cardio-vascular disorders
* Major neurologic disorders
* Major ocular disorders
* Morphine in pre-operative period

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2004-01-31 (Actual); Primary Completion 2005-07-31 (Actual); Study Completion 2005-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie COLOMBANI, MD, Principal Investigator — Institut Bergonié
Locations (1):
- Institut Bergonié - Centre Régional de Luttre Contre le Cancer de Bordeaux et du Sud Ouest, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Ketamine Arm: Anesthetic induction: Ketamine at 0.15 mg/kg is added to the "Reference protocol".
  Anesthetic maintenance: Ketamine at 2 mg/kg/min is added to the "Reference protocol".
  Ketamine
- Reference Arm: Induction and anesthetic maintenance without ketamine (reference arm / saline solution)
  Saline solution
Period: Overall Study
Arm/Group | Ketamine Arm | Reference Arm
Started | 115 | 115
Completed | 109 | 104
Not Completed | 6 | 11
Not completed — Withdrawal by Subject | 3 | 2
Not completed — absence of lymph node dissection after intraoperative frozen section of the specimen | 3 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ketamine Arm | Reference Arm | Total
Number analyzed (Participants) | 109 | 104 | 213
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.4 (12.3) | 58.8 (11.4) | 58 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 109 | 104 | 213
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  France | 109 | 104 | 213

OUTCOME MEASURES:

1. Primary Outcome: Morphine Consumption (First 48 Post-operative Hours)
Description: Number of participants with at least one consumption of morphine within 48 hours following surgery.
Time Frame: within 48 hours following surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Ketamine Arm | Reference Arm
Number analyzed (Participants) | 109 | 104
Participants | 79 | 77

2. Secondary Outcome: Post-operative Pain
Description: Count of participants with post-operative pain. Pain was measured using a Visual Analog Rating Scale (VAS), ranging from 0 (no pain) to 10 (pain).
  A VAS score >= 4 wwas considered as "Pain". A VAS sore <4 was considered as "No pain".
Time Frame: 48 hours after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Ketamine Arm | Reference Arm
Number analyzed (Participants) | 109 | 104
Participants
  No pain (VAS < 4) | 106 | 102
  Pain (VAS >= 4) | 3 | 2

ADVERSE EVENTS:
Time Frame: 6 months after surgery
Arm/Group | Ketamine Arm | Reference Arm
All-Cause Mortality (participants affected / at risk) | 0/109 | 0/104
Serious Adverse Events (participants affected / at risk) | 0/109 | 0/104
Other Adverse Events (participants affected / at risk) | 20/109 | 14/104
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ketamine Arm (N=109) | Reference Arm (N=104)
Nausea (Gastrointestinal disorders) | 8 (8) | 8 (8)
Vomiting NOS (Gastrointestinal disorders) | 12 (12) | 12 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes